CLINICAL TRIAL: NCT06771128
Title: Ginkgo Biloba Versus Desmopressin in Treatment of Children With Monosymptomatic Nocturnal Enuresis: A Randomized Prospective Study
Brief Title: Ginkgo Biloba vs Desmopressin in Treatment of Children With Monosymptomatic Nocturnal Enuresis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ammar Fathi Mohamed AlOrabi, Doctor, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ginkgo Biloba vs Desmopressin
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-09

CONDITIONS: Nocturnal Enuresis in Children; Desmopressin; Monosymptomatic Nocturnal Enuresis
Keywords: monosymptomatic nocturnal enuresis; nocturnal enuresis; desmopressin; Ginkgo Biloba
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Ginkgo Extract; Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ginkgo Biloba group (Experimental): Patients in this group receive Ginkgo Biloba oral tablet.
  Interventions: Drug: Ginkgo Biloba oral tablet; Drug: Desmopressin like Placebo
- Desmopressin group (Active Comparator): Patients in this group receive Desmopressin oral tablets.
  Interventions: Drug: Desmopressin Acetate 0.2 mg Tablets; Drug: Ginkgo Biloba like Placebo
- Combination group (Experimental): Patients in this group receive both Ginkgo Biloba and desmopressin oral tablets.
  Interventions: Drug: Ginkgo Biloba oral tablet; Drug: Desmopressin Acetate 0.2 mg Tablets
- Placebo group (Placebo Comparator): Patients in this group receive Placebo oral tablet.
  Interventions: Drug: Ginkgo Biloba like Placebo; Drug: Desmopressin like Placebo

INTERVENTIONS:
Drug: Ginkgo Biloba oral tablet — patients receive Ginkgo Biloba oral tablet 120 mg once daily
  Arms: Combination group; Ginkgo Biloba group
Drug: Desmopressin Acetate 0.2 mg Tablets — patient receives desmopressin 0.2 mg oral tablet once daily
  Arms: Combination group; Desmopressin group
Drug: Ginkgo Biloba like Placebo — patients receive Ginkgo Biloba like Placebo oral tablet once daily
  Arms: Desmopressin group; Placebo group
Drug: Desmopressin like Placebo — patients receive Desmopressin like Placebo oral tablet once daily
  Arms: Ginkgo Biloba group; Placebo group

SUMMARY:
the efficacy of Ginkgo Biloba versus desmopressin in treatment of children with monosymptomatic nocturnal enuresis

DETAILED DESCRIPTION:
Bedwetting among children is a common disorder, affecting 30% at age 4, 10% at age 6, 3% at age 12, and 1% at age. Untreated, the spontaneous cure rate is about 15% a year. Treatment is dominated by two approaches, enuresis alarm and drugs.

Treatment with drugs has largely been focused on tricyclic antidepressants especially imipramine or, more recently, antidiuretic agents such as desmopressin. For imipramine the proportion of total remission is 10-50% during treatment and a long term cure in 5-40%. However, numerous reports of side effects, some lethal, have led to a decline in its use.

One of theory of nocturnal enuresis is deep sleep in children, this the main cornerstone in using Alarm as line of management.

On the other hand drugs used in re-habitation of sleep rhythm seems to be with great benefits in management as GINKGO BILOBA.

Ginkgo biloba leave extract is among the most widely sold herbal dietary supplements in the United States. Its purported biological effects include: scavenging free radical; lowering oxidative stress; reducing neural damages, reducing platelets aggregation; anti-inflammation; anti-tumor activities; anti-aging, and improve night sleep rhythm.

the aim of this study is to evaluate the effect of Ginkgo Biloba versus desmopressin in treatment of children with monosymptomatic nocturnal enuresis.

ELIGIBILITY:
Inclusion Criteria:

* all children with monosymptomatic nocturnal enuresis.

Exclusion Criteria:

* children with day and night wetting.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 398 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Night wetting frequency | 1, 3 months
  Night wetting frequency is measured by the number of wet nights per week.

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia Faculty of Medicine, Shebin El-Kom, Menoufia, Egypt